CLINICAL TRIAL: NCT04994392
Title: Intra-Operative Complication Assessment and Reporting With Universal Standards: Surgeons, Anesthesiologists, and Nurses Survey
Brief Title: Intra-Operative Complication Assessment and Reporting With Universal Standards: Survey
Acronym: ICARUS-S
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Giovanni Cacciamani, Assistant Professor of Urology (research), University of Southern California
Other Study IDs: UP-21-00473
Record Dates: First submitted 2021-07-10; First posted 2021-08-06 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Intraoperative Complications; Surgery--Complications; Surgery; Surgical Procedure, Unspecified
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perioperative complications, especially intraoperative adverse events (iAEs), carry significant potential for long-term sequelae in a patient's postoperative course. Without consistent and homogenous reporting, these events represent a substantial gap in contemporary surgical literature and clinical practice. By definition, an iAE is any unplanned incident related to a surgical intervention occurring between skin incision and skin closure.

Despite the availability of multiple intraoperative classification systems, the reporting of intraoperative adverse events remains exceedingly rare. Further, while most studies report postoperative adverse events, only a fraction of surgical publications report intraoperative complications as outcomes of interest. Many reasons could be related to this dearth in iAE reporting, ranging from a lack of clear iAE definitions to a fear of litigation. Broadly speaking, iAEs are negative outcomes, which, on the whole, epitomize a paradoxically well-documented bias in the literature.

The investigators performed an umbrella review and meta-analysis of prior systematic reviews of complication reporting in a number of key urologic surgical domains. The investigators have since worked with academic surgeons to produce a set of iAE reporting guidelines known as the Intraoperative Complication Assessment and Reporting with Universal Standards (ICARUS) Guidelines. These reporting criteria were developed using the reporting guidelines using the framework outlined by the EQUATOR Network (Enhancing the QUAlity and Transparency Of health Research; www.equator-network.org/).

As part of a prospective effort to evaluate the utility of these new guidelines, the investigators are performing a study of surgeons, anesthesiologists,s and nurses perceptions regarding iAE reporting and the global applicability of the new iAE reporting guidelines.

In part one of this study, a series of survey questions will be used to better elucidate surgeon perceptions underlying the contemporary deficit in iAE reporting. In part two of this study, a set of assessments to representatives within various surgical specialties to assess the global applicability of the newly developed iAE reporting guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Documented understanding, willingness, and agreement to participate in this study
2. Males and females; age 18 or older
3. Must be either English speaking or fluent with English medical terminology
4. Currently or formerly practicing surgeon or proceduralist, regardless of the domain

Exclusion Criteria:

1. Activity restrictions that limit one's ability to engage in online survey

1. Adults not competent to consent
2. Minors, human fetuses, neonates
3. Prisoners/Detainees

The sample size of the survey is calculated as reported by Taherdoost, Hamed et al. Determining Sample Size; How to Calculate Survey Sample Size (2017). International Journal of Economics and Management Systems, Vol. 2, 2017, considering the worldwide surgeons and anesthesiologists population (n. 1,853,842) accordingly to the most recent WHO Surgical workforce Census (https://apps.who.int/gho/data/view.main.HRSWF),with a 95% Level and 2% marginal error.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study team will identify corresponding authors who have published articles at any point during 2019-2021 in key American and European scientific surgical journals. The study team plans to email up to 1500 authors from each of these journals - though, many of these journals will not likely have substantially fewer corresponding authors. Specifically, these journals will be associated with one or more of the following specialties:
  * Anesthesiology
  * Interventional Radiology
  * Interventional Cardiology
  * Nursing
  * Cardiothoracic surgery
  * Colon and rectal surgery
  * General surgery
  * Gynecologic oncology
  * Gynecology and obstetrics
  * Neurological surgery
  * Ophthalmologic surgery
  * Oral and maxillofacial surgery
  * Orthopaedic surgery
  * Otorhinolaryngology
  * Plastic surgery
  * Urology
  * Vascular Surgery
Sampling Method: Non-Probability Sample
Enrollment: 4821 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Global perception of intraoperative adverse event reporting | July 30th 2021 till September 30th 2021
  A series of 5-point Likert scale assessments relating to surgeon perception of intraoperative adverse assessment as it related to the following domains: reporting habits, practical considerations, clinical and quality improvement utility, emotional response, and perceived consequences. The questions do not include any validated questionnaires or psychometric evaluations. Descriptive statistical assessment of responses.
Global applicability of the ICARUS reporting criteria | July 30th 2021 till September 30th 2021
  Determination of global applicability (clinical utility and quality improvement utility) of the ICARUS reporting criteria as determined by subjective 5-point Likert scale assessments. Outcomes to be assessed by percent agreement and interrater consistency.

SECONDARY OUTCOMES:
Specialty specific perception of intraoperative adverse event reporting | July 30th 2021 till September 30th 2021
  A series of 5-point Likert scale assessments relating to surgeon perception of intraoperative adverse assessment as it related to the following domains: reporting habits, practical considerations, clinical and quality improvement utility, emotional response, and perceived consequences. The questions do not include any validated questionnaires or psychometric evaluations. Descriptive statistical assessment of responses.
Specialty-specific applicability of ICARUS guidelines | July 30th 2021 till September 30th 2021
  Determination of specialty specific applicability (clinical utility and quality improvement utility) of the ICARUS reporting criteria as determined by subjective 5-point Likert scale assessments. Outcomes to be assessed by percent agreement and interrater consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni E Cacciamani, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Background] Taherdoost, Hamed, Determining Sample Size; How to Calculate Survey Sample Size (2017). International Journal of Economics and Management Systems, Vol. 2, 2017, Available at SSRN: https://ssrn.com/abstract=3224205
- [Result] Biyani CS, Pecanka J, Roupret M, Jensen JB, Mitropoulos D. Intraoperative Adverse Incident Classification (EAUiaiC) by the European Association of Urology ad hoc Complications Guidelines Panel. Eur Urol. 2020 May;77(5):601-610. doi: 10.1016/j.eururo.2019.11.015. Epub 2019 Nov 29. PMID 31787430
- [Result] Rosenthal R, Hoffmann H, Clavien PA, Bucher HC, Dell-Kuster S. Definition and Classification of Intraoperative Complications (CLASSIC): Delphi Study and Pilot Evaluation. World J Surg. 2015 Jul;39(7):1663-71. doi: 10.1007/s00268-015-3003-y. PMID 25665678
- [Result] Kaafarani HM, Mavros MN, Hwabejire J, Fagenholz P, Yeh DD, Demoya M, King DR, Alam HB, Chang Y, Hutter M, Antonelli D, Gervasini A, Velmahos GC. Derivation and validation of a novel severity classification for intraoperative adverse events. J Am Coll Surg. 2014 Jun;218(6):1120-8. doi: 10.1016/j.jamcollsurg.2013.12.060. Epub 2014 Feb 28. PMID 24702887
- [Result] Kazaryan AM, Rosok BI, Edwin B. Morbidity assessment in surgery: refinement proposal based on a concept of perioperative adverse events. ISRN Surg. 2013 May 16;2013:625093. doi: 10.1155/2013/625093. Print 2013. PMID 23762627
- [Result] Han K, Bohnen JD, Peponis T, Martinez M, Nandan A, Yeh DD, Lee J, Demoya M, Velmahos G, Kaafarani HMA. The Surgeon as the Second Victim? Results of the Boston Intraoperative Adverse Events Surgeons' Attitude (BISA) Study. J Am Coll Surg. 2017 Jun;224(6):1048-1056. doi: 10.1016/j.jamcollsurg.2016.12.039. Epub 2017 Jan 16. PMID 28093300
- [Result] Cacciamani GE, Maas M, Nassiri N, Ortega D, Gill K, Dell'Oglio P, Thalmann GN, Heidenreich A, Eastham JA, Evans CP, Karnes RJ, De Castro Abreu AL, Briganti A, Artibani W, Gill I, Montorsi F. Impact of Pelvic Lymph Node Dissection and Its Extent on Perioperative Morbidity in Patients Undergoing Radical Prostatectomy for Prostate Cancer: A Comprehensive Systematic Review and Meta-analysis. Eur Urol Oncol. 2021 Apr;4(2):134-149. doi: 10.1016/j.euo.2021.02.001. Epub 2021 Mar 6. PMID 33745687
- [Result] Cacciamani GE, Medina LG, Tafuri A, Gill T, Baccaglini W, Blasic V, Glina FPA, De Castro Abreu AL, Sotelo R, Gill IS, Artibani W. Impact of Implementation of Standardized Criteria in the Assessment of Complication Reporting After Robotic Partial Nephrectomy: A Systematic Review. Eur Urol Focus. 2020 May 15;6(3):513-517. doi: 10.1016/j.euf.2018.12.004. Epub 2018 Dec 23. PMID 30587445